CLINICAL TRIAL: NCT06608901
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamic Effects of REGN7544, an Antagonist Monoclonal Antibody to NPR1, in Patients With Sepsis-Induced Hypotension
Brief Title: A Study of REGN7544 for the Treatment in Adult Patients With Sepsis-Induced Hypotension
Acronym: ESTELLA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R7544-SIH-2435; 2024-514946-35-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Sepsis-Induced Hypotension
Keywords: Natriuretic Peptide Receptor 1 (NPR1); Low Blood Pressure
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- REGN7544 (Experimental)
  Interventions: Drug: REGN7544
- Placebo (PB) (Placebo Comparator)
  Interventions: Drug: PB

INTERVENTIONS:
Drug: REGN7544 — Administered per the protocol
  Arms: REGN7544
Drug: PB — Administered per the protocol
  Arms: Placebo (PB)

SUMMARY:
This study is researching an experimental drug called REGN7544 (called "study drug"). The study is focused on adult patients (18 to 85 years) hospitalized due to a serious infection (called "sepsis") and receiving standard-of-care medications for low blood pressure (called "vasopressors") due to sepsis.

The aim of the study is to see how safe, tolerable, and effective the study drug is by observing the effects on blood pressure and the total amount of vasopressor dose received during the stay in the hospital.

The study is looking at several other research questions, including:

* How the study drug changes the blood pressure and the amount of intravenous (IV) fluids given to participants with low blood pressure due to sepsis
* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Proven or suspected infection defined as administration or planned administration of antimicrobial therapy within the screening period
2. Sepsis-induced hypotension that has not responded to Intravenous (IV) fluids, receiving 1 or 2 vasopressors and maintaining a Mean Arterial Pressure (MAP) of ≥ 65 mm Hg for at least 2 consecutive hours immediately prior to randomization, as defined in the protocol

Key Exclusion Criteria:

1. Unable to obtain informed consent by participant or Legally Authorized Representative (LAR)
2. Clinical status requires vasopressor and/or Blood Pressure (BP) management inconsistent with the study protocol
3. Primary cause of hypotension suspected to be due to non-sepsis cause (eg, hemorrhage, burns, or cardiogenic shock), including shock after cardiac arrest
4. Ejection fraction <20% in the most recent known echocardiogram
5. Acute coronary syndrome based on clinical symptoms and/or electrocardiogram (ECG) during hospitalization
6. History of hospitalization due to heart failure, myocardial infarction, stroke, clinically significant ventricular arrhythmia, transient ischemic attack, or unstable angina within the preceding 3 months
7. Any prior diagnosis of severe pulmonary hypertension, as defined in the protocol
8. Receiving 3 or more vasopressors or exceeding the maximal combined dose as defined in the protocol, during the screening period or at the time of study drug administration
9. Received bone marrow transplant during the preceding 6 months or chemotherapy during the preceding 30 days for lymphoma or leukemia

NOTE: Other Protocol-Defined Inclusion-Exclusion Criteria Apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-07-23 (Estimated); Study Completion 2026-10-19 (Estimated)

PRIMARY OUTCOMES:
Cumulative vasopressor dose | Through 72 Hours

SECONDARY OUTCOMES:
Occurrence of Common Terminology Criteria for Adverse Events (CTCAE) grade 3 and higher Treatment-Emergent Adverse Events (TEAEs) | Through 90 Days
Time-weighted average Mean Arterial Pressure (MAP) | Baseline Over 4 Hours
Change in MAP | Baseline, At 4 Hours
Proportion of surviving participants free of vasopressor(s) | At 24, 48 and 72 Hours
Cumulative net fluid balance | Through 72 Hours
Cumulative urine output | Through 72 Hours
Cumulative fluid intake | Through 72 Hours
Concentrations of REGN7544 in serum | Through 90 Days
Incidence of Anti-Drug Antibodies (ADA) to REGN7544 | Through 90 Days
Magnitude of ADA to REGN7544 | Through 90 Days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (29):
- United States (16):
  - University of Arizona, Tucson, Arizona
  - Yale University, New Haven, Connecticut
  - Emory University Hospital, Atlanta, Georgia
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Harvard Medical School - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - New York University Langone Health Brooklyn Hospital, Brooklyn, New York
  - Bellevue Hospital, New York, New York
  - New York University Langone Health Tisch-Kimmel Hospital, New York, New York
  - Montefiore Medical Center - Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Atrium Health, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - MUSC SCTR Research Nexus Clinic and Lab, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Intermountain Medical Center - Murray (Pulmonary Medicine), Murray, Utah
- France (13):
  - Centre Hospitalier Regional Universaitaire de Tours (CHRU de Tours), Tours, Centre-Val de Loire
  - CHU Dupuytren, Limoges, Nouvelle-Aquitaine
  - Centre Hospitalier Le Mans, Le Mans, Pays de la Loire Region
  - Centre Hospitalier Departemental (CHD) Vendee, La Roche-sur-Yon, Vendee
  - Centre Hospitalier Universitaire Angers, Angers
  - Raymond Poincare University Hospital, Garches
  - Paris-Saclay University Hospitals, Le Kremlin-Bicêtre
  - CHU Nantes, Nantes
  - Centre Hospitalier Universitaire d'Orleans, Orléans
  - CHU de Reims Hopital Robert Debre, Reims
  - Hopitaux Universitaires de Strasbourg, Strasbourg
  - Hopital Nord Franche Comte, Trévenans
  - Hopital Cochin, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/